CLINICAL TRIAL: NCT06581055
Title: A Retrospective Study to Describe Real-World Treatment Patterns and Clinical Outcomes Among Patients With Myelodysplastic Syndromes Who Discontinued Treatment With Luspatercept or Epoetin Alfa and the COMMANDS Trial
Brief Title: A Retrospective Study to Describe Real-World Treatment Patterns and Clinical Outcomes Among Patients With Myelodysplastic Syndromes
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1083
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Myelodysplastic syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept; Epoetin Alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Luspatercept: Adult participants treated with and discontinued Luspatercept treatment while enrolled in the COMMANDS trial (NCT03682536).
  Interventions: Drug: Luspatercept
- Epoetin alfa: Adult participants treated with and discontinued Epoetin alfa treatment while enrolled in the COMMANDS trial (NCT03682536).
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Luspatercept — As per COMMANDS Trial (NCT03682536) study protocol
  Groups: Luspatercept
Drug: Epoetin Alfa — As per COMMANDS Trial (NCT03682536) study protocol
  Groups: Epoetin alfa

SUMMARY:
This study aims to collect real-world data on treatment patterns and clinical outcomes for participants who discontinued Luspatercept or epoetin alfa treatment and discontinued the COMMANDS trial (NCT03682536) utilizing existing data from patient medical records.

ELIGIBILITY:
Inclusion Criteria:

* Participant was enrolled in and discontinued the COMMANDS trial.
* Participant was treated with either luspatercept or epoetin alfa and discontinued treatment while enrolled in the COMMANDS trial.
* Participant Patient provides informed consent (only where applicable or required by local regulations).

Exclusion Criteria:

• There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult participants with myelodysplastic syndromes who were enrolled in the COMMANDS trial (NCT03682536) and discontinued Luspatercept or Epoetin alfa treatment and discontinued the COMMANDS trial.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Participant treatment patterns: Type of treatment received | Up to 24 months
Participant treatment patterns: Duration of treatment received | Up to 24 months
Participant treatment patterns: Dosage of treatment received | Up to 24 months
Participant treatment patterns: Dosing route of treatment administration | Up to 24 months
Participant treatment patterns: Reason for treatment administration | Up to 24 months
Participant treatment patterns: Time to next line of therapy (LoT) | Up to 24 months
Participant treatment patterns: Reason for treatment discontinuation | Up to 24 months
Participant treatment patterns: Type of concomitant medications received | Up to 24 months
Participant treatment patterns: Start and end dates of concomitant medications received | Up to 24 months

SECONDARY OUTCOMES:
Participant clinical outcomes: Number of units of red blood cell transfusions received | Up to 24 months
Participant clinical outcomes: Red blood cell transfusion burden (RBC-TB) category | Up to 24 months
  Category 1: Transfusion dependent (at least 4 units of red blood cell (RBC) with 8 weeks for hemoglobin (Hb) <9g/dL) Category 2: Transfusion independence (<4 units of RBC with 8 weeks for Hb <9 g/dL)
Participant clinical outcomes: Red blood cell transfusion burden (RBC-TB) category per International Working Group (IWG) 2018 | Up to 24 months
  IWG 2028 criteria:
  1. Non-transfused (0 Red Blood Cells [RBC] in 16 weeks)
  2. Low-transfusion burden (3-7 RBCs in 16 weeks in at least 2 transfusion episodes, maximum 3 in 8 weeks)
  3. High-transfusion burden (≥8 RBCs in 16 week, ≥4 in 8 weeks)
Participant clinical outcomes: Blood test results | Up to 24 months
Participant clinical outcomes: Number of participants that progressed to acute myeloid leukemia (AML) status | Up to 24 months
Number of participants that progressed to high-risk myelodysplastic syndromes (MDS) | Up to 24 months
Participant clinical outcomes: Participant survival status | Up to 24 months
Participant clinical outcomes: Date and primary cause of death | Up to 24 months
Participant clinical characteristics | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- National Taiwan University Hospital (NTUH), Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts